CLINICAL TRIAL: NCT02134366
Title: A Phase III, Randomized, Open Label, Single Center, Study on the Effects of Treatment of Epilepsia Partialis Continua With Clobazam Compared to Treatment With or in Addition to Lorazepam and/or Clonazepam
Brief Title: Clobazam Use in Epilepsia Partialis Continua - Pilot Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment Issues - Lack of target population
Sponsor: The Cooper Health System (Other)
Collaborators: Lundbeck LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: EPC-1
Record Dates: First submitted 2014-05-06; First posted 2014-05-09 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Epilepsia Partialis Continua; Kojewnikov's Epilepsy; Epilepsy
Keywords: Epilepsia Partialis Continua; Kojewnikov's Epilepsy; Epilepsy; Clobazam; Focal Motor Epilepsy; Partial Motor Seizure
MeSH Terms: conditions — Epilepsia Partialis Continua; Epilepsy; Epilepsy, Partial, Motor | interventions — Clobazam; Clonazepam; Lorazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clobazam (Experimental): Subjects who are assigned the clobazam treatment group will receive a 10mg loading dose followed by a maintenance dose of 5-25 mg bid starting 12 hrs after the loading dose. If subjects are found to have failed to respond to treatment with clobazam, the physician investigator has the ability to either start another AED or increase the dose of clobazam depending on the clinical situation. Subjects still being treated with clobazam at discharge will be given a 30 day supply of clobazam.
  Interventions: Drug: Clobazam; Drug: Clonazepam; Drug: Lorazepam
- Clonazepam (Active Comparator): Subjects who are assigned to the clonazepam treatment group will receive a dose of 1-2mg clonazepam dose tid. Following the initial treatment if a physician investigator determines that the subject's treatment has failed, the investigator has the option of treating the subject with clobazam at which point the individuals would be treated in the same method as those originally assigned to the clobazam treatment group.
  Interventions: Drug: Clobazam; Drug: Clonazepam; Drug: Lorazepam
- Lorazepam (Active Comparator): Subjects who are assigned to the lorazepam treatment group will receive a 1-2mg dose of lorazepam qid. Following the initial treatment if a physician investigator determines that the subject's treatment has failed, the investigator has the option of treating the subject with clobazam at which point the individuals would be treated in the same method as those originally assigned to the clobazam treatment group.
  Interventions: Drug: Clobazam; Drug: Clonazepam; Drug: Lorazepam

INTERVENTIONS:
Drug: Clobazam — Comparison of AED use in Epilepsia Partialis Continua
  Other Names: Onfi; Frisium; Urbanol
Drug: Clonazepam — Comparison of AED use in Epilepsia Partialis Continua
  Other Names: Klonopin
Drug: Lorazepam — Comparison of AED use in Epilepsia Partialis Continua
  Other Names: Ativan; Orfidal

SUMMARY:
The purpose of this study is to evaluate whether clobazam, brand name Onf®, is more effective as an adjunctive or monotherapy in terminating Epilepsia Partialis Continua (EPC) than either lorazepam and/or clonazepam.

DETAILED DESCRIPTION:
First approved in the United States in 2011 for use in treating Lennox-Gastaut syndrome, clobazam is the only 1, 5-benzodiazepine that is currently approved for clinical use in the United States. In previous clinical trials clobazam has been shown to have a greater efficacy and produce fewer side effects in individuals when it's adverse event profile is compared to the traditional 1,4-benzodiazepines such as diazepam, lorazepam, and clonazepam. As a benzodiazepine, clobazam has been found to have anticonvulsant properties, and structural differences as a 1,5-benzodiazepines that appear to have a broader spectrum of anticonvulsant activity than those found in 1,4-benzodiazepines. In previous reports, clobazam has been seen to be effective in ether terminating or reducing both EPC in particular and partial status epilepticus.

ELIGIBILITY:
Inclusion Criteria:

•≥ to 18 yrs of age

•Diagnosis of EPC by a Neurologist

Exclusion Criteria:

* Previous exposure to clobazam prior to presentation
* Seizure generalization
* Patients who are intubated and on IV sedation such as Versed®, Propofol or Presedex®.
* Female subjects who are pregnant and/or breast-feeding
* Subject has an unstable and/or serious or psychiatric illness
* Subject has an unstable and/or serious medical illness
* Subject has any of the following but not limited to conditions:

  * A life threatening medical condition
  * Severe sepsis or septic shock
  * Severe Renal impairment
  * Severe Hepatic impairment
  * Sleep apnea
  * Narrow angle glaucoma
  * Severe respiratory insufficiency
  * Myasthenia gravis
  * Metastatic cancer
  * Organ failure
  * Severe progressive nervous system disease
  * A clinically significant EKG abnormality that would be affected by and/or affect the patient's participation in the trial
* Subject has active suicidal ideation at Screening and Baseline visits
* Subject has a history of suicidal thoughts or behaviors, which would be indicated by a positive response to questions 4 and/or 5 on the CSSR-S. Exclusionary actions include but are not limited to:

  * Previous intent to act on suicidal ideation with a specific plan
  * Previous preparatory acts or behavior
  * A previous actual attempt, interrupted attempt or aborted suicide attempt
* Subject has a history of alcohol and/or substance abuse in the previous 12 months, or the subject is unable to refrain from alcohol and/or substance abuse during the study.
* Subject admits to present illicit drug use or has a positive drug screen
* Subject is currently enrolled in or has been enrolled in any clinical trial within the past 30 days
* Subject has a known allergy to any component of the study medication(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Time (measured in minutes) to onset of seizure freedom | Within 7 days
Reduction of seizure frequency/minute | Within 7 days

SECONDARY OUTCOMES:
Mental status preservation off sedating anticonvulsants as measured by the MoCA© scale | Within 37 days
Ambulatory function as measured by the Hauser Ambulation Index | Within 37 days

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Carran, MD, Principal Investigator — Cooper University Health System
Locations (1):
- Cooper Universtiy Hospital, Camden, New Jersey, United States